CLINICAL TRIAL: NCT05162287
Title: Psychosocial Distress, Levels of Personality Functioning, and Social Withdrawal in a Child and Adolescent Psychiatric Acute Inpatient Population
Brief Title: Child and Adolescent Psychiatric Personality Structure
Acronym: CAPPS
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Johannes Boettcher, Dipl.-Psych., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 2021-100618-BO-FF
Record Dates: First submitted 2021-11-10; First posted 2021-12-17 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Personality Disorders; Social Withdrawal of Childhood or Adolescence; Psychosocial Impairment
Keywords: acute adolescent psychiatric units
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who are treated in the acute ward of the child and adolescent psychiatry: All children and adolescents aged 12 to 18 years who are treated in the acute ward of the Department of Child and Adolescent Psychiatry, Psychotherapy and Psychosomatics at the University Medical Center Hamburg-Eppendorf are recruited.

SUMMARY:
The study plan outlined here represents an investigation of instruments on the patients treated in the acute ward of child and adolescent psychiatry at the University Medical Center Hamburg Eppendorf (UKE). The psychosocial burden of the affected children and adolescents is evident due to the severity of the disorders leading to specific admission. The psychosocial burden can be defined as "psychological, social, or school-occupational functional impairment [...] that has arisen as a consequence of a mental disorder, a specific developmental disorder, or an intellectual impairment". The current research project aims to survey the severity of psychosocial distress, personality functioning impairment, and social withdrawal. A better knowledge of these factors may contribute to a more suitable, specialized treatment offer on the acute ward in the medium term.

DETAILED DESCRIPTION:
Children and adolescents who receive inpatient psychiatric treatment are counted among the most impaired in society. In addition to the usually very severe mental disorders, the patient:s often have psychosocial risk factors and traumatic life events in their history. As demand for psychiatric-psychotherapeutic care increases, many inpatient services have been driven to reduce costs, while parallel pressures to measure outcomes and effectiveness have increased. The call for evidence-based practice underscores the need to use valid and reliable measurement tools to capture changes in symptoms and functionality during short-term interventions and their effectiveness. Measuring this change allows for the evaluation of the interventions as a whole and identifying areas for improvement. Acute care units are a particular type of inpatient setting. The main goal of treatment is to stabilize the patient:s by reducing acute psychiatric symptoms, suicide risk, and danger to others. The challenge of care for this target group is to do justice to heterogeneous initial situations and offer customized help for each child and adolescent. The use of instruments to record psychosocial stress and personality disorders increases the chance that at least some of those affected can be prevented from developing a chronic course and thus long-term psychosocial impairment utilizing tailored interventions.

ELIGIBILITY:
Inclusion criteria

* Patients treated in the acute ward of the Department of Child and Adolescent Psychiatry, Psychotherapy, and Psychosomatics at the University Medical Center Hamburg-Eppendorf
* Patients with a principal diagnosis of a psychiatric disorder (ICD-10-GM-2016: F10 - F90).
* Patients under 18 years of age.

Exclusion criteria

* Patients with organic, including symptomatic mental disorders (F00 - F09)
* Dementia / cognitive impairment (IQ < 70)
* lack of German language skills
* severe visual or hearing impairment (uncorrected).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Clinical study participants for the diagnostic study are patients between the ages of 12 and 17 who are undergoing treatment for a psychiatric illness in the acute care unit of the Child and Adolescent Psychiatry Department at the University Medical Center Hamburg-Eppendorf.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Psychosocial distress | 7 minutes
  HoNOSCA-D (Dölitzsch et al., 2020; von Wyl et al., 2017) The Health of the Nation Outcomes Scales for Children and Adolescents (HoNOSCA) is a questionnaire assessing psychosocial distress in children and adolescents. The 13-item instrument is a viable tool for differentiating the severity and social functioning of those with mental illness and can be used as a meaningful outcome instrument. It parallels a clinician's external assessment with a self-assessment.
Psychosocial distress | 3 minutes
  CGAS (Shaffer et al., 1983): adapted from the Global Assessment Scale for adults, the Children's Global Assessment Scale (CGAS) assesses functioning aimed at children and adolescents aged 6-17 years. The child or adolescent receives a single score ranging from 1 to 100 based on a clinician's assessment of several aspects of the child's psychological and social functioning. The score can be placed in one of ten categories ranging from "extremely impaired" to "very good"

SECONDARY OUTCOMES:
Level of personality functioning | 5 minutes
  SEFP (Falkai & Wittchen, 2015b): The level of personality functioning is dimensionally classified in the alternative DSM-5-PS model using the Level of Personality Functioning Scale. Criterion A is based on a normative functioning model of personality, from which there can be defined deviations, divided into four degrees of severity, regarding identity, self-control, empathy, and closeness. The SEFP is determined by an assessment by a clinician.
Level of personality functioning | 10 minutes
  LoPF-Q 12-18 (Goth et al., 2018b): The Levels of Personality Functioning 12-18 Questionnaire (LoPF-Q 12-18) instrument assesses self-report impairments in personality functioning in the four domains of identity, self-control, empathy, and closeness in children and adolescents between the ages of 12 and 18. The test allows a dimensional differentiation between healthy and impaired personality functions, which are associated with a high risk of an existing personality disorder.
Social withdrawal | 3 minutes
  YSR/11-18 (Döpfner et al., 2014): Social withdrawal is measured with nine items from the Youth Self-Report 11-18 (YSR/11-18), the social withdrawal subscale. The YSR is a widely used 112-item self-report scale of emotional and behavioral problems developed for children and adolescents ages 11 to 18. Items can be rated on a 3-point scale, where 0=not at all; 1=sometimes or not at all; and 2=always or often true in the past 6 months.
Social withdrawal | 2 minutes
  3-item Loneliness Scale (Klein et al., 2021): Social withdrawal is also measured by the 3-item Loneliness Scale. The scale is an economic measure derived from the R-UCLA Loneliness Scale (Russell et al., 1980) that captures basic aspects of loneliness: A sense of isolation, disconnectedness, and not belonging. Items are rated on 5-point Likert scales (0=never, 1=sometimes, 2=sometimes, 3=often, 4=very often). Responses are summed for a total score ranging from 0 to 12, with higher scores indicating higher levels of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Boettcher, M.Sc., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychotherapy and Psychosomatics; Carola Bindt, PD Dr., Study Director — Department of Child and Adolescent Psychiatry, Psychotherapy and Psychosomatics; Ursula Völker, Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychotherapy and Psychosomatics
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided if there will be a plan to make IPD available.

REFERENCES:
- [Background] Remschmidt, H., Schmidt, M. H., & Poustka, F. (2017). Multiaxiales Klassifikationsschema für psychische Störungen des Kindes- und Jugendalters nach ICD-10 (7th ed.). Hogrefe AG.
- [Background] Kronstrom K, Ellila H, Kuosmanen L, Kaljonen A, Sourander A. Changes in the clinical features of child and adolescent psychiatric inpatients: a nationwide time-trend study from Finland. Nord J Psychiatry. 2016 Aug;70(6):436-41. doi: 10.3109/08039488.2016.1149617. Epub 2016 Mar 22. PMID 27002640
- [Background] Hall CL, Moldavsky M, Taylor J, Sayal K, Marriott M, Batty MJ, Pass S, Hollis C. Implementation of routine outcome measurement in child and adolescent mental health services in the United Kingdom: a critical perspective. Eur Child Adolesc Psychiatry. 2014 Apr;23(4):239-42. doi: 10.1007/s00787-013-0454-2. Epub 2013 Jul 30. No abstract available. PMID 23896764
- [Background] Tharayil PR, Sigrid J, Morgan R, Freeman K. Examining Outcomes of Acute Psychiatric Hospitalization among Children. Soc Work Ment Health. 2012;10(3):205-232. doi: 10.1080/15332985.2011.628602. PMID 23946699
- [Background] Yuan JM. HoNOSCA in an adolescent psychiatric inpatient unit: an exploration of outcome measures. Psychiatr Danub. 2015 Sep;27 Suppl 1:S357-63. PMID 26417796
- [Background] Schmeck, K., & Schlüter-Müller, S. (2021). Identitätsentwicklung als Fokus von psychodynamischer Kinder- und Jugendpsychotherapie. PDP - Psychodynamische Psychotherapie, 20(1), 28-39. https://doi.org/10.21706/pdp-20-1-28
- [Background] Goth K, Birkholzer M, Schmeck K. Assessment of Personality Functioning in Adolescents With the LoPF-Q 12-18 Self-Report Questionnaire. J Pers Assess. 2018 Nov-Dec;100(6):680-690. doi: 10.1080/00223891.2018.1489258. PMID 30907712
- [Background] Fonagy P, Speranza M, Luyten P, Kaess M, Hessels C, Bohus M. ESCAP Expert Article: borderline personality disorder in adolescence: an expert research review with implications for clinical practice. Eur Child Adolesc Psychiatry. 2015 Nov;24(11):1307-20. doi: 10.1007/s00787-015-0751-z. Epub 2015 Aug 14. PMID 26271454
- [Background] Chanen A, Sharp C, Hoffman P; Global Alliance for Prevention and Early Intervention for Borderline Personality Disorder. Prevention and early intervention for borderline personality disorder: a novel public health priority. World Psychiatry. 2017 Jun;16(2):215-216. doi: 10.1002/wps.20429. No abstract available. PMID 28498598